CLINICAL TRIAL: NCT00188409
Title: Pneumothorax Following CT-Guided Lung Biopsy: Is There a Role for the Post Biopsy CT in Patient Management
Brief Title: Pneumothorax Post CT Lung Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0122
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2005-09

CONDITIONS: Lung Nodules

INTERVENTIONS:
Procedure: CT scan

SUMMARY:
A CT scan is performed after a lung biopsy in order to detect a Pneumothorax. We postulate that CT is more useful than chest radiography

ELIGIBILITY:
Inclusion Criteria:

* all patients having a lung biopsy

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2002-02; Study Completion 2004-02

PRIMARY OUTCOMES:
detection of pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: narinder paul, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada